CLINICAL TRIAL: NCT03386149
Title: Clinical Research on the Efficacy and Safety of Bosinji on LBP and Radiculopathy by HIVD of L-spine; A Multicenter, Randomized, Controlled, Clinical Trial
Brief Title: Clinical Research on the Efficacy of Bosinji on Herniated Intervertebral Disc of Lumbar Spine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Kyung Hee University Hospital at Gangdong (Other); DongGuk University (Other); Daegu Korean Medicine Hospital of Daegu Haany University (Other)
Responsible Party: Principal Investigator, Byung-Kwan Seo, Principal Investigator, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KHNMCOH 2017-08-002
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Lumbar Disc Herniation
Keywords: Herniated Intervertebral Disc of Lumbar Spine; Low Back Pain; Radiculopathy; Bosinji; Herbal Medicine
MeSH Terms: conditions — Intervertebral Disc Displacement; Low Back Pain; Radiculopathy | interventions — loxoprofen; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): In the experimental group, 2.5g of Bosinji granule (Tsmura Co., Tokyo, Japan) will be orally administered three times a day at 30 minutes after the meal for 6 weeks. During the same period, acupuncture treatment on 20 predefined acupoints will be conducted once a week.
  Interventions: Drug: Bosinji; Procedure: Acupuncture
- Control Group (Active Comparator): In the control group, Loxonine tab. (loxoprofen 60mg, Dong Wha Pharm Co., Ltd, Seoul, Korea) will be orally administered three times a day at 30 minutes after the meal for 6 weeks. During the same period, acupuncture treatment on 20 predefined acupoints will be conducted once a week.
  Interventions: Drug: Loxonine tab.; Procedure: Acupuncture

INTERVENTIONS:
Drug: Bosinji — Product name : Bosinji Granule Manufacturer : Tsumura & Co. Ingredient : Bosinji granule 2.5g (Bosinji extract 1.523g)
  Bosinji extract is composed of following proportion of ingredient
  * Rehmannia Root 1.7g
  * Achyranthes Root 1.0g
  * Cornus Fruit 1.0g
  * Dioscorea Rhizome 1.0g
  * Psyllium Husk 1.0g
  * Alisma Rhizome 1.0g
  * Hoelen 1.0g
  * Moutan Root Bark 1.0g
  * Cinnamon Bark 0.3g
  * Pulvis Aconiti Tuberis Purificatum 0.3g
  Other Names: Ucha-Shinki-Hwan
  Arms: Experimental Group
Drug: Loxonine tab. — Product name : Loxonine tab. Manufacturer : Dong Wha Pharm. Co., Ltd Ingredient : Loxoprofen Sodium 68.1mg (Loxoprofen 60mg)
  Other Names: Loxoprofen
  Arms: Control Group
Procedure: Acupuncture — Acupuncture treatment will be performed on 20 predefined acupoint using 0.25mm x 40mm acupuncture needle. The time for needle retaining is 15 minutes.
  1. Both EX-B2 of herniated intervertebral disc level, its upper level and its lower level (6 acupoints)
  2. Both side BL24, BL25, BL26, EX-B7, BL28 (10 acupoints)
  3. Symptomatic side GB30, GB34, BL57, ST36 (4 acupoints)

SUMMARY:
This randomized controlled clinical trial is designed to evaluate the efficacy and safety of Bosinji on low back pain and radiating pain of lumbar herniated intervertebral disc (L-HIVD) by assessing pain, function, and quality of life.

DETAILED DESCRIPTION:
Seventy-four patients between the ages of 19 and 70 with L-HIVD will be recruited by eligibility criteria and randomly allocated to the experimental group and the control group. In the experimental group, 2.5g of Bosinji granule (Tsumura & Co., Tokyo, Japan) will be orally administered three times a day at 30 minutes after the meal for 6 weeks. In the control group, Loxonine tab. (loxoprofen 60mg, Dong Wha Pharm Co., Ltd, Seoul, Korea) will be orally administered in the same usage and period with the experimental group. In addition, both group will receive the same acupuncture treatment on 20 acupoints once a week for 6 weeks. 100 mm visual analogue scale (VAS) for low back pain will be assessed as a primary outcome at baseline and treatment end. Also, 100mm VAS for radiating pain, Oswestry disability index (ODI), Rolland Morris disability questionnaire (RMDQ), EQ-5D-5L and global perceived effect (GPE), Deficiency Syndrome of Kidney Index (DSKI) will be measured as secondary outcomes at baseline, 3 weeks after screening, treatment end (6 weeks, primary endpoint) and follow-up sessions (10 weeks).

ELIGIBILITY:
Inclusion Criteria:

1. Men or women aged over 19 years
2. Radiating pain matched with severer abnormality than bulging shown by CT or MRI on lumbar spine
3. low back pain between 40 and 80 point on 100mm pain visual analogue scale
4. Volunteers who agree to participate and sign the Informed Consent Form, following a detailedexplanation of clinical trials

Exclusion Criteria:

1. Congenital abnormalities or surgical history on lumbar regions
2. Red flag signs that may be suspected of cauda equina syndrome, such as bladder and bowel dysfunction or saddle anesthesia
3. Tumor, fracture or infection in lumbar regions
4. Injection treatment on lumbar regions within 1 week
5. Psychiatric disorder currently undergoing treatment such as depression or schizophrenia
6. Liver function abnormality (AST or ALT over 2times normal range)
7. Renal fuction abnormaility (Serum creatinine > 2.0㎎/㎗)
8. Other diseases that could affect or interfere with therapeutic outcomes, including severe gastrointestinal disease, cardiovascular disease, hypertension, diabetes, renal disease, liver disease or thyroid disorder
9. Contraindication of NSAIDs including intercurrent disease, hypersensitivity reaction or other medication
10. Inappropriate condition for acupuncture due to skin disease or hemostatic disorder (PT INR > 2.0 or taking anticoagulant)
11. Women who is pregnant, breastfeeding or having pregnancy plan
12. Other inappropriate condition for herbal medicine treatment
13. participation in other clinical trial with 1 month

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-12-28 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Change from Baseline 100mm Pain Visual Analogue Scale (VAS) for low back pain at Week 6 | Week 0 (Baseline), Week 3, Week 6 (Primary end point, Treatment end), Week 10 (F/U)
  Measurement instrument for subjective pain

SECONDARY OUTCOMES:
100mm Pain Visual Analogue Scale (VAS) for radiating pain | Week 0 (Baseline), Week 3, Week 6 (Primary end point, Treatment end), Week 10 (F/U)
  Measurement instrument for subjective pain
Oswestry Disability Index (ODI) | Week 0 (Baseline), Week 3, Week 6 (Primary end point, Treatment end), Week 10 (F/U)
  Validated questionnaire for disability of low back pain
EuroQol-5 dimensions-5 level (EQ-5D-5L) | Week 0 (Baseline), Week 3, Week 6 (Primary end point, Treatment end), Week 10 (F/U)
  Standardized instrument for generic health status
Roland-Morris Disability Questionnaire (RMDQ) | Week 0 (Baseline), Week 3, Week 6 (Primary end point, Treatment end), Week 10 (F/U)
  Health status measure for low back pain
Global Perceived Effect (GPE) | Week 3, Week 6 (Primary end point, Treatment end), Week 10 (F/U)
  Assessment of change in the patient's chief complaint
Deficiency Syndrome of Kidney Index (DSKI) | Week 0 (Baseline), Week 6 (Primary end point, Treatment end)
  Questionnaire for assessing symptoms related to deficiency syndrome of kidney

CONTACTS AND LOCATIONS:
Overall Officials: Byung-Kwan Seo, PhD., KMD, Principal Investigator — Kyunghee University Medical Center
Locations (4):
- South Korea (4):
  - Dongguk University Bundang Oriental Hospital, Seongnam-si, Gyeonggi-do
  - Daegu Korean Medicine Hospital of Daegu Haany University, Daegu
  - Kyunghee University Medical Center, Seoul
  - Kyung Hee University Hospital at Gangdong, Seoul

REFERENCES:
- [Derived] Goo B, Kim JH, Kim EJ, Nam D, Lee HJ, Kim JS, Park YC, Baek YH, Nam SS, Seo BK. Clinical research on the effectiveness and safety of Uchasingihwan for low back pain with radiculopathy caused by herniated intervertebral disc of the lumbar spine: A multicenter, randomized, controlled equivalence trial. Integr Med Res. 2024 Dec;13(4):101090. doi: 10.1016/j.imr.2024.101090. Epub 2024 Sep 30. PMID 39640075
- [Derived] Goo B, Kim SJ, Kim EJ, Nam D, Lee HJ, Kim JS, Park YC, Baek YH, Nam SS, Seo BK. Clinical research on the efficacy and safety of Bosinji for low back pain with radiculopathy caused by herniated intervertebral disc of the lumbar spine: A protocol for a multicenter, randomized, controlled equivalence trial. Medicine (Baltimore). 2018 Dec;97(50):e13684. doi: 10.1097/MD.0000000000013684. PMID 30558079